CLINICAL TRIAL: NCT05138575
Title: SGLT2i and KNO3 in HFpEF - The SAK HFpEF Trial
Acronym: SAK
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Payman Zamani, MD, Principle Investigator, University of Pennsylvania
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 849401
Record Dates: First submitted 2021-11-03; First posted 2021-12-01 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Heart Failure With Preserved Ejection Fraction
MeSH Terms: interventions — empagliflozin; Potassium Chloride; potassium nitrate

STUDY DESIGN:
Intervention Model Description: 3 interventions will be randomized and administered in a double-blind fashion
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All personnel will be masked except for the IDS pharmacist dispensing the drugs.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Empagliflozin + Potassium Chloride (KCl) (Active Comparator): Empagliflozin (10 mg daily) + Potassium Chloride (6 mmol three times daily)
  Active arm will be 6 weeks in duration followed by a 2 week washout period.
  Interventions: Drug: Empagliflozin + Potassium Chloride
- Empagliflozin + Potassium Nitrate (KNO3) (Active Comparator): Empagliflozin (10 mg daily) + Potassium Nitrate (6 mmol three times daily)
  Active arm will be 6 weeks in duration followed by a 2 week washout period.
  Interventions: Drug: Empagliflozin + Potassium Nitrate
- Potassium Chloride (KCl) + Placebo for Empa (Placebo Comparator): Potassium Chloride (6 mmol three times daily) + Placebo for Empagliflozin
  Placebo arm will be 6 weeks in duration followed by a 2 week washout period.
  Interventions: Drug: Potassium Chloride + Placebo for Empagliflozin

INTERVENTIONS:
Drug: Empagliflozin + Potassium Chloride — Empagliflozin is the active intervention that may improve mitochondrial function and energy fuel metabolism in skeletal muscle.
  KCl is an active control.
  Other Names: Jardiance + KCl
  Arms: Empagliflozin + Potassium Chloride (KCl)
Drug: Empagliflozin + Potassium Nitrate — Empagliflozin + KNO3 is the active intervention that may improve mitochondrial function and energy fuel metabolism in skeletal muscle, as well as increase skeletal muscle perfusion during exercise.
  Other Names: Jardiance + KNO3
  Arms: Empagliflozin + Potassium Nitrate (KNO3)
Drug: Potassium Chloride + Placebo for Empagliflozin — Active control.
  Other Names: KCl + Placebo
  Arms: Potassium Chloride (KCl) + Placebo for Empa

SUMMARY:
This study will test whether pharmacologic agents that may improve mitochondrial function and energy fuel metabolism [Empagliflozin (Empa)], with and without additional supplements that increase perfusion and fatty acid oxidation [Potassium Nitrate (KNO3)], improve submaximal exercise endurance and skeletal muscle oxidative phosphorylation capacity (SkM OxPhos) in participants with Heart Failure with Preserved Ejection Fraction (HFpEF).

DETAILED DESCRIPTION:
This study will test whether Empagliflozin (Empa), with and without Potassium Nitrate (KNO3), improves submaximal exercise endurance, skeletal muscle oxidative phosphorylation capacity (SkM OxPhos), intramuscular perfusion, and changes in the skeletal muscle metabolome, proteome, and respiration in participants with Heart Failure with Preserved Ejection Fraction (HFpEF).

ELIGIBILITY:
Inclusion:

1. NYHA Class II-III symptoms 2. Left ventricular ejection fraction >= 50% 3. Stable medical condition for at least 2 weeks, as per investigator judgment 4. Prior or current evidence for elevated filling pressures, as evidenced by at least one of the following:

a. Mitral early (E)/septal tissue annular (e') velocity ratio > 8, in the context of a septal e' velocity <=7 cm/s or a lateral e' <= 10 cm/s, in addition to one of the following: i. Large left atrium (LA volume index > 34 mL/m2) ii. Chronic loop diuretic use for control of symptoms iii. Elevated natriuretic peptides within the past year (e.g., NTproBNP > 125 pg/mL in sinus rhythm or > 375 pg/mL if in atrial fibrillation) b. Mitral E/e' ratio > 14 at rest or during exercise c. Elevated invasively-determined filling pressures previously (resting left ventricular end-diastolic pressure >= 16 mm Hg or pulmonary capillary wedge pressure >= 15 mmHg; or PCWP/LVEDP >= 25 mmHg with exercise) d. Prior episode of acute heart failure requiring IV diuretics

Exclusion Criteria:

1. Age <18 years old
2. Pregnancy: Women of childbearing potential will undergo a urine pregnancy test during the screening visit.
3. Treatment with organic nitrates or phosphodiesterase inhibitors that cannot be interrupted
4. Uncontrolled atrial fibrillation, as defined by a resting atrial fibrillation heart rate > 100 beats per minute at the time of the baseline assessment
5. Hemoglobin < 10 g/dL
6. Subject inability/unwillingness to exercise
7. Moderate or greater left sided valvular disease (mitral regurgitation, aortic stenosis, aortic regurgitation), mild or greater mitral stenosis, severe right-sided valvular disease
8. Known hypertrophic, infiltrative, or inflammatory cardiomyopathy
9. Clinically significant pericardial disease, as per investigator judgment
10. Current angina due to clinically significant epicardial coronary disease, as per investigator judgment
11. Acute coronary syndrome or coronary intervention within the past 2 months
12. Primary pulmonary artery hypertension (WHO Group 1 Pulmonary Arterial Hypertension)
13. Clinically significant lung disease as defined by: Chronic Obstructive Pulmonary Disease Stage III or greater GOLD criteria (FEV1<50%), treatment with oral steroids within the past 6 months for an exacerbation of obstructive lung disease, current use of supplemental oxygen aside from nocturnal oxygen for the treatment of obstructive sleep apnea.

    - Desaturation to <90% on the baseline maximal effort cardiopulmonary exercise test will also be grounds for exclusion
14. Clinically-significant ischemia, as per investigator's judgement, on stress testing without either (1) subsequent revascularization, (2) an angiogram demonstrating the absence of clinically significant epicardial coronary artery disease, as per investigator judgment; (3) a follow-up 'negative' stress test, particularly when using a more specific technique (i.e., a negative perfusion imaging test following a 'positive' ECG stress test)

    - Exercise-induced regional wall motion abnormalities on the echocardiographic assessment during the baseline maximal effort cardiopulmonary exercise test will also be exclusionary
15. Left ventricular ejection fraction < 45% on a prior echocardiogram or cardiac MRI, unless the reduced LVEF occurred within the context of an uncontrolled supraventricular arrhythmia, with return of a normal ejection fraction following treatment of the arrhythmia
16. Significant liver disease impacting synthetic function or volume control (ALT/AST > 3x ULN, Albumin < 3.0 g/dL)
17. eGFR < 30 mL/min/1.73m2.
18. Methemoglobin > 5%
19. Serum potassium > 5.0 mEq/L on baseline testing
20. Type I Diabetes
21. History of ketoacidosis
22. Current use of, or prior intolerance to, an SGLT2i
23. Ongoing maintenance of a 'Ketogenic Diet' (low carbohydrate, high fat)
24. Allergy to beets
25. Severe right ventricular dysfunction
26. Baseline resting seated systolic blood pressure > 180 mmHg or < 100 mmHg
27. Persistently low or high seated blood pressure or orthostatic blood pressure response to the transition from supine to standing (>20 mmHg reduction in systolic blood pressure 2-3 minutes after standing, or a fall in SBP to < 90 mmHg) at the baseline visit
28. Active participation in another study that utilizes an investigational agent (observational studies/registries allowed)
29. Any condition that, in the opinion of the investigator, may interfere with the completion/performance of the study. This may include comorbid or psychiatric conditions that may impede successful completion of the protocol, or logistical concerns (e.g., inability to travel to the exercise unit).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2022-01-24 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Submaximal Exercise Endurance | Week 6
  Time to exhaustion while exercising at 75% peak workload

SECONDARY OUTCOMES:
Intramuscular Perfusion | Week 6
  MRI assessment of skeletal muscle perfusion
VO2 Kinetics | Week 6
  Assess the impact of interventions on the kinetics of oxygen consumption (VO2 kinetics) during exercise and recovery. "On" and "Off" kinetics will be modeled during the submaximal exercise transient.
VO2 Efficiency | Week 6
  Assess the impact of interventions on the efficiency of oxygen consumed above basal metabolic rate compared to total work performed
Vasodilatory Reserve | Week 6
  Percent change in systemic vascular resistance (SVR) at baseline vs SVR at 4 minutes of exercise at end of each intervention period
Venous Substrate Concentration | Week 6
  Change in venous substrate concentrations at time of fatigue at end of each intervention period
Respiratory Exchange Ratio | Week 6
  Change in RER at 4 minutes of exercise at end of each intervention period
KCCQ Overall Summary Score | Week 6
  Assess impact of interventions on quality of life based on Kansas City Cardiomyopathy Questionnaire overall summary score
Ambulatory Physical Activity | Week 6
  Use actigraphy to document the average steps per day taken during the final week of each interventional period
Muscle Tissue Respirometry | Week 6
  Measure tissue rates of substrate metabolism and mitochondrial content
Muscle Proteome | Week 6
  Measure relative abundances of proteins related to fatty acid and ketone oxidation as well as proteins related to mitochondrial biogenesis.
Muscle Metabolome | Week 6
  Perform targeted quantitative metabolomics to assess changes in substrate metabolism
Skeletal Muscle Oxidative Capacity | Week 6
  MRI assessment of skeletal muscle oxidative phosphorylation capacity
Arteriovenous O2 content difference | Week 6
  quotient of VO2 to cardiac output
Peak VO2 during Submaximal Exercise | Week 6
  Assess the impact of interventions on the peak oxygen consumption achieved during submaximal exercise

OTHER OUTCOMES:
Intramyocardial Filling Pressure | Week 6
  Assess impact of interventions on intramyocardial filling pressures during submaximal exercise

CONTACTS AND LOCATIONS:
Overall Officials: Payman Zamani, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania Health System, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Study participant research data, which is for purposes of statistical analysis and scientific reporting, will be maintained indefinitely in an electronic database. This will not include the participant's contact or identifying information. Rather, individual participants and their research data will be identified by a unique study identification number. The study data entry and study management systems used by clinical sites and by the research staff will be secured and password protected. At the end of the study, all study databases will be de-identified and archived.
  If any data or samples are shared with collaborators at UPenn or elsewhere, only de-identified samples/data will be given, without any linking information.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-28): https://cdn.clinicaltrials.gov/large-docs/75/NCT05138575/Prot_SAP_000.pdf
  • Informed Consent Form (2021-09-28): https://cdn.clinicaltrials.gov/large-docs/75/NCT05138575/ICF_001.pdf